CLINICAL TRIAL: NCT00315341
Title: Starting Treatment With Agonist Replacement Therapies (START)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Walter Ling, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0027; U10DA013045 (NIH)
Record Dates: First submitted 2006-04-16; First posted 2006-04-18 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Opiate-related Disorders
MeSH Terms: interventions — Buprenorphine, Naloxone Drug Combination; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine/Nx (Experimental): For the BUP/NX group, all participants will receive up to 16 mg BUP/4 mg NX on day 1 and up to 32 mg BUP/8 mg NX on day 2. It is recommended that dose changes be made in 2 to 8 mg buprenorphine increments, with the range of allowable daily doses between 2 mg and 32 mg starting on day 3 and thereafter according to clinical impression and depending upon the participant's clinical need. Investigators are encouraged to dose adequately to decrease craving and to obtain negative urine toxicology specimens.
  Interventions: Drug: Buprenorphine/naloxone
- Methadone (Active Comparator): For the MET group, all participants will receive a maximum of 30 mg for the first dose and a maximum of 40 mg on Day 1. It is recommended that participants receive a dose on day 2 that is 10 mg higher than their total day 1 dose, and a dose on day 3 that is 10 mg higher than their total day 2 dose, unless, in the clinical judgment of the physician, a slower induction is needed. Doses will be adjusted on Day 4 and thereafter according to clinical impression and depending upon the participant's clinical need with no specific upper limit. Investigators are encouraged to dose adequately to decrease craving and to obtain negative urine toxicology specimens.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Participants receive up to 16 mg BUP/4 mg NX on day 1 and up to 32 mg BUP/8 mg NX on day 2. It is recommended that dose changes be made in 2 to 8 mg increments, with the range of allowable daily doses between 2 mg and 32 mg starting on day 3 and thereafter according to clinical impression and depending upon the participant's clinical need.
  Arms: Buprenorphine/Nx
Drug: Methadone — Participants will receive a maximum of 30 mg for the first dose and a maximum of 40 mg on Day 1. It is recommended that participants receive a dose on day 2 that is 10 mg higher than their total day 1 dose, and a dose on day 3 that is 10 mg higher than their total day 2 dose, unless, in the clinical judgment of the physician, a slower induction is needed. Doses will be adjusted on Day 4 and thereafter according to clinical impression and depending upon the participant's clinical need with no specific upper limit.
  Arms: Methadone

SUMMARY:
The Food and Drug Administration (FDA) has requested a study comparing buprenorphine/naloxone (BUP/NX) and methadone (MET) on indices of hepatic safety.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, Phase 4 study to assess the changes in liver enzymes related to treatment with buprenorphine/naloxone (BUP/NX) and methadone (MET) in participants entering opioid agonist treatment. Randomization will be stratified, within site, according to normal versus abnormal screening liver function tests. Participants meeting entry criteria will be dosed for 24 weeks during the active phase of the study with assessment of liver function at weeks 1, 2, 4, 8, 12, 16, 20, 24 and with follow-up assessments at week 32. Clinicians will be encouraged to treat with adequate doses of BUP/NX and MET.

ELIGIBILITY:
Inclusion Criteria:

1. Were age 18 years or older,
2. Met DSM-IV-TR criteria for opioid dependence,
3. Were in good general health, or, in case of a medical/psychiatric condition requiring ongoing treatment, were under the care of a physician willing to continue participant's medical management and cooperate with study physicians,
4. For female participants, use of one of the following acceptable methods of birth control:

   1. oral contraceptives
   2. barrier (diaphragm or condom) with spermicide
   3. IUD
   4. intrauterine progesterone contraceptive system
   5. levonorgestrel implant
   6. medroxyprogesterone acetate contraceptive injection
   7. contraceptive transdermal patch
   8. hormonal vaginal contraceptive ring
   9. surgical sterilization
   10. complete abstinence from sexual intercourse
5. Able to read and verbalize understanding of the study and voluntarily sign study informed consent form.

Exclusion Criteria:

1. ALT or AST values > 5 times the upper limit of normal as per testing laboratory range criteria,
2. ALP values >3 times the upper limit of normal per testing laboratory criteria,
3. Any documented past or present history of ascites, presence of esophageal or gastric varices, hepatic encephalopathy or other signs of significant liver disease as indicated by a Model for Endstage Liver Disease score (Kamath et al., 2001) of ≥11,
4. Total bilirubin > 2.0 mg/dl (participants with documented Gilbert's syndrome were not excluded based on this criterion),
5. Prothrombin time more than 3 seconds prolonged,
6. Albumin level less than 2.5 g/dl,
7. Any cardiopathy or risk factor listed below without evidence of a normal ECG* with report performed within 6 months prior to first study medication dose,

   1. Congestive heart failure
   2. Left ventricular hypertrophy
   3. Bradycardia
   4. Hereditary QT prolongation
   5. Uncorrected electrolyte imbalance
   6. Concomitant medications that are known to have a risk of QT interval prolongation; refer to Appendix D for a list of medications.

   Note: The list was not all-inclusive.

   *An ECG was abnormal if one or more of the following occurred:

   Significant ST segment abnormalities:
   * ST segment elevations in two or more continuous leads of > 0.1 mV
   * ST segment depression of greater than 1 mm that are flat or down-sloping at 80 msec after the J point ST segment abnormalities identified as "non-specific" are acceptable. If a potential participant's ECG indicated ST segment elevations or depression consistent with ischemia, the physician obtained a medical history of cardiac symptoms and referred the participant for evaluation.

   Conduction abnormalities:
   * Mobitz II 2nd degree or 3rd degree heart block
   * Atrial fibrillation, atrial flutter, or any non-sinus tachyarrhythmia
   * Three or more consecutive ectopic ventricular complexes at a rate of > 100 per minute.
   * QTc greater than 450 msec in men and 480 msec in women

   Repolarization abnormalities:

   • Acute medical condition that would make participation, in the opinion of the study physician, medically hazardous (e.g., unstable pancreatic, cardiovascular or renal disease, significant anemia)
8. Known allergy or sensitivity to BUP, naloxone or MET or to any of the inactive ingredients in the study medications (including lactose, mannitol, cornstarch, povidone K30, citric acid, sodium citrate, FD&C Yellow No.6 color, magnesium stearate, Acesulfame K sweetener)
9. Known diagnosis of acute psychosis, severe depression or imminent suicide risk as determined via clinical interview by study physician or surrogates
10. DSM-IV diagnosis of dependence on alcohol requiring immediate medical attention.
11. DSM-IV diagnosis of dependence on benzodiazepines requiring immediate medical attention
12. DSM-IV diagnosis of dependence on other depressants, or stimulants requiring immediate medical attention
13. Participation in an investigational drug study within the past 30 days
14. Treatment with MET, BUP/NX, or BUP for more than 15 of the past 30 days (illicit use of these medications is allowed)
15. Pending legal action that could prohibit study participation
16. Unable or unwilling to comply with study requirements
17. Unable or unwilling to remain in the local area for duration of treatment
18. Poor venous access such that venipuncture could not be accomplished from a vein in an extremity during eligibility
19. Pregnant or lactating (females only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1269 (Actual)
Dates: Start 2006-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — University of California, Los Angeles; Andrew Saxon, M.D., Principal Investigator — University of Washington
Locations (9):
- United States (9):
  - Matrix Institute, Los Angeles, California
  - Bi-Valley Medical Clinic INC., Sacramento, California
  - BAART; Turk Street Clinic, San Francisco, California
  - Hartford Dispensary, Hartford, Connecticut
  - CT Counseling Centers, Waterbury, Connecticut
  - Addiction Research & Treatment Corp, Brooklyn, New York
  - CODA-Research, Portland, Oregon
  - NET Steps, Philadelphia, Pennsylvania
  - Evergreen Treatment Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saxon AJ, Ling W, Hillhouse M, Thomas C, Hasson A, Ang A, Doraimani G, Tasissa G, Lokhnygina Y, Leimberger J, Bruce RD, McCarthy J, Wiest K, McLaughlin P, Bilangi R, Cohen A, Woody G, Jacobs P. Buprenorphine/Naloxone and methadone effects on laboratory indices of liver health: a randomized trial. Drug Alcohol Depend. 2013 Feb 1;128(1-2):71-6. doi: 10.1016/j.drugalcdep.2012.08.002. Epub 2012 Aug 22. PMID 22921476
- [Derived] Brandt L, Odom GJ, Hu MC, Castro C, Balise RR; CTN-0094 Team. Empirically contrasting urine drug screening-based opioid use disorder treatment outcome definitions. Addiction. 2024 Jul;119(7):1289-1300. doi: 10.1111/add.16494. Epub 2024 Apr 14. PMID 38616571
- [Derived] Wang K, Shafique S, Xiao D, Walter SM, Liu Y, Piamjariyakul U, Xie C. Repeated measures analysis of opioid use disorder treatment on clinical opiate withdrawal scale in a randomized clinical trial: sex differences. J Addict Dis. 2024 Jan-Mar;42(1):33-44. doi: 10.1080/10550887.2022.2131957. Epub 2023 Jan 19. PMID 36655851
- [Derived] Nielsen S, Tse WC, Larance B. Opioid agonist treatment for people who are dependent on pharmaceutical opioids. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD011117. doi: 10.1002/14651858.CD011117.pub3. PMID 36063082
- [Derived] Nwabueze C, Elom H, Liu S, Walter SM, Sha Z, Acevedo P, Liu Y, Su BB, Xu C, Piamjariyakul U, Wang K. Gender differences in the associations of multiple psychiatric and chronic conditions with major depressive disorder among patients with opioid use disorder. J Addict Dis. 2022 Apr-Jun;40(2):168-178. doi: 10.1080/10550887.2021.1957639. Epub 2021 Jul 30. PMID 34328394
- [Derived] Crist RC, Li J, Doyle GA, Gilbert A, Dechairo BM, Berrettini WH. Pharmacogenetic analysis of opioid dependence treatment dose and dropout rate. Am J Drug Alcohol Abuse. 2018;44(4):431-440. doi: 10.1080/00952990.2017.1420795. Epub 2018 Jan 15. PMID 29333880
- [Derived] Woody GE, Bruce D, Korthuis PT, Chhatre S, Poole S, Hillhouse M, Jacobs P, Sorensen J, Saxon AJ, Metzger D, Ling W. HIV risk reduction with buprenorphine-naloxone or methadone: findings from a randomized trial. J Acquir Immune Defic Syndr. 2014 Jul 1;66(3):288-93. doi: 10.1097/QAI.0000000000000165. PMID 24751432
- [Derived] Hser YI, Saxon AJ, Huang D, Hasson A, Thomas C, Hillhouse M, Jacobs P, Teruya C, McLaughlin P, Wiest K, Cohen A, Ling W. Treatment retention among patients randomized to buprenorphine/naloxone compared to methadone in a multi-site trial. Addiction. 2014 Jan;109(1):79-87. doi: 10.1111/add.12333. Epub 2013 Oct 9. PMID 23961726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Methadone clinics in California, Oregon, Washington, Pennsylvania, New York, and Connecticut
Groups:
- Buprenorphine/Nx: Participants received medication for 24 weeks in the active phase of the study. The mean dose of buprenorphine was 22.3 mg. Blood samples for measurement of liver function were taken at baseline and at Weeks 1, 2, 4 8, 12, 16, 20, and 24 with follow-up at Week 32.
- Methadone: The mean dose of methadone was 93.2 mg.
Period: Overall Study
Arm/Group | Buprenorphine/Nx | Methadone
Started | 740 | 529
Completed | 340 | 391
Not Completed | 400 | 138

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine/Nx | Methadone | Total
Number analyzed (Participants) | 740 | 529 | 1269
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.2) | 37.3 (10.9) | 37.4 (11.1)
Gender [Count of Participants; unit: Participants]
  Female | 238 | 170 | 408
  Male | 502 | 359 | 861

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Safety
Description: Participants were categorized according liver transaminase (ALT, AST) levels in blood comparing the baseline sample to any and all subsequent samples in the following manner:
  A: both ALT and AST started at less than or equal to two times the ULN and remained at two times or less ULN throughout the study
  B: either ALT or AST started at less than or equal to 2 x ULN and at any point in study exceeded 2 x ULN
  C: Either ALT or AST started > 2 x ULN, decreased (both ALT and AST) to < 2 x ULN, and remained < 2 x ULN
  D: Either ALT or AST started > 2 x ULN and remained above 2 x ULN throughout the study
Time Frame: 24 Weeks
Population: evaluable subjects stayed in treatment for 24 weeks and gave at least 4 blood samples for liver function tests during the treatment period
Measure: Number; unit: participants
Arm/Group | Buprenorphine/Nx | Methadone
Number analyzed (Participants) | 340 | 391
participants
  ALT - A (low, stays low) | 278 | 318
  ALT - B (low, goes high) | 41 | 62
  ALT - C (high, goes low, stays low) | 4 | 1
  ALT - D (high, stays high) | 17 | 10
  AST - A (low, stay low) | 291 | 328
  AST - B (low, goes high) | 37 | 54
  AST - C (high, goes low, stays low) | 3 | 1
  AST - D (high, stays high) | 9 | 8
Statistical Analysis 1: Comparison: Buprenorphine/Nx vs Methadone; categorized changes in ALT/AST from BL:(1)BL transaminases(both ALT/AST)≤2X upper limit of normal(ULN)& remained at this level;(2)BL transaminases ≤2X ULN(either ALT/AST)but increased(either ALT/AST)above this level at any time;(3)BL transaminases >2X ULN(either ALT/AST)& decreased and remained at ≤2X ULN(both ALT/AST);(4)BL transaminases(both ALT/AST)>2X ULN &remained at this level(both ALT/AST);(5)BL transaminases >2X ULN(either ALT/AST)& increased 2X above this level ever(either ALT/AST); Test type: Superiority or Other; p < 0.05, shift table analyses

ADVERSE EVENTS:
Time Frame: Adverse events (medical and/or psychiatric) assessment will initiate with participant randomization and will continue through 30 days post last dose of study medication administered. Study staff should contact each participant 30 days after study completion and/or discontinuation of study medication to follow-up on any adverse events continuing at study end and to determine whether the participant experienced any adverse events within the 30 days after discontinuing study medication.
Description: All AEs reported during the course of the study requiring medical attention will be reported to a study physician immediately. A study physician may then meet any participants for whom additional follow-up or AE assessment is indicated. The type of AE, severity of the AE and the relationship of the AE to the study treatments will be assessed by appropriately trained medical personnel and recorded on an AE CRF, according to the procedures described in Section 14.2.
Arm/Group | Buprenorphine/Nx | Methadone
Serious Adverse Events (participants affected / at risk) | 38/727 | 45/520
Other Adverse Events (participants affected / at risk) | 530/727 | 442/520
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Nx (N=727) | Methadone (N=520)
death (Investigations) | 3 (3) | 1 (1)
life-threatening (Investigations) | 3 (3) | 3 (3)
hospitalization (Investigations) | 38 (41) | 45 (50)
disability (Investigations) | 0 (0) | 4 (4)
congenital anomaly (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Nx (N=727) | Methadone (N=520)
alanine aminotransferase increased (Investigations) | 81 (104) | 70 (94)
aspartate aminotransferase increased (Investigations) | 70 (78) | 63 (87)
gamma glutamyltransferase increased (Investigations) | 47 (54) | 57 (71)
weight increased (Investigations) | 10 (10) | 26 (26)
nasopharyngitis (Infections and infestations) | 119 (147) | 117 (165)
influenza (Infections and infestations) | 35 (38) | 34 (37)
upper respiratory tract infection (Infections and infestations) | 32 (38) | 26 (30)
toothache (Gastrointestinal disorders) | 49 (60) | 55 (72)
constipation (Gastrointestinal disorders) | 49 (52) | 47 (51)
vomiting (Gastrointestinal disorders) | 28 (28) | 30 (36)
injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 134 (238) | 124 (218)
nervous system disorders (Nervous system disorders) | 154 (246) | 106 (151)
headache (Nervous system disorders) | 102 (132) | 54 (72)
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 135 (208) | 98 (136)
back pain (Musculoskeletal and connective tissue disorders) | 50 (56) | 37 (43)
psychiatric disorders (Psychiatric disorders) | 114 (162) | 89 (129)
general disorders and administration site conditions (General disorders) | 79 (99) | 83 (162)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 75 (92) | 75 (98)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 (13) | 38 (44)
respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 82 (105) | 64 (80)
investigations (Investigations) | 215 (564) | 214 (619)
infections and infestations (Infections and infestations) | 281 (470) | 249 (466)
gastrointestinal disorders (Gastrointestinal disorders) | 196 (311) | 174 (291)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No